CLINICAL TRIAL: NCT07329972
Title: A Phase 1, Open-label, Randomized, Crossover Study to Evaluate the Effect of Food and Proton Pump Inhibitor on the Pharmacokinetics of ZN-A-1041 Tablet(s) in Healthy Participants
Brief Title: A Study to Evaluate the Effect of Food and Proton Pump Inhibitor on the Pharmacokinetics of ZN-A-1041 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GP46367
Record Dates: First submitted 2025-11-20; First posted 2026-01-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Sequence 1 (Experimental)
  Interventions: Drug: ZN-A-1041 Formulation 1; Drug: Rabeprazole
- Sequence 2 (Experimental)
  Interventions: Drug: ZN-A-1041 Formulation 1; Drug: Rabeprazole
- Sequence 3 (Experimental)
  Interventions: Drug: ZN-A-1041 Formulation 1; Drug: Rabeprazole
- Sequence 4 (Experimental)
  Interventions: Drug: ZN-A-1041 Formulation 1; Drug: Rabeprazole
- Sequence 5 (Experimental)
  Interventions: Drug: ZN-A-1041 Formulation 2; Drug: Rabeprazole
- Sequence 6 (Experimental)
  Interventions: Drug: ZN-A-1041 Formulation 2; Drug: Rabeprazole
- Sequence 7 (Experimental)
  Interventions: Drug: ZN-A-1041 Formulation 2; Drug: Rabeprazole
- Sequence 8 (Experimental)
  Interventions: Drug: ZN-A-1041 Formulation 2; Drug: Rabeprazole

INTERVENTIONS:
Drug: ZN-A-1041 Formulation 1 — Participants will receive a single dose of ZN-A-1041 Formulation 1 on each specified treatment.
  Arms: Sequence 1; Sequence 2; Sequence 3; Sequence 4
Drug: ZN-A-1041 Formulation 2 — Participants will receive a single dose of ZN-A-1041 Formulation 2 on each specified treatment.
  Arms: Sequence 5; Sequence 6; Sequence 7; Sequence 8
Drug: Rabeprazole — Participants will receive an oral administration of rabeprazole twice daily (BID) on days 9, 10, 15, and 16 and a single dose on Days 11 and 17.

SUMMARY:
This study is a phase 1, open-label, randomized, four-period crossover study to evaluate the effect of food and rabeprazole on the ZN-A-1041 tablet formulation in healthy male and female participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within the range of 18 to 32 kg/m2, inclusive
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs, as determined by the investigator, at Screening and Check-in, as applicable
* Clinical laboratory evaluations (including chemistry panel, CBC, and UA with complete microscopic analysis) within the normal reference ranges for the certified test laboratory at Screening and Check-in
* Negative test for selected drugs of abuse at Screening and Check-in (includes alcohol)
* Negative hepatitis panel (hepatitis B surface antigen, hepatitis B core antibody, hepatitis B surface antibody [unless consistent with vaccination or immunity due to natural infection], and hepatitis C virus antibody) and negative HIV antibody screens
* For women of childbearing potential: agreement to remain abstinent or use contraception
* For men: agreement to remain abstinent or use contraceptive methods, and agreement to refrain from donating sperm
* Negative screening test for latent Mycobacterium tuberculosis infection
* Able to swallow and retain multiple tablets without chewing or crushing
* Able to consume the high-fat meal within the protocol-specified time period and willing to consume 100% of the high-fat meal
* Able to fast for 8 hours prior to dosing

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), neurological, or psychiatric disorder, as determined by the investigator
* History or concurrent clinically significant hemorrhagic, bleeding abnormalities, as determined by the investigator
* Personal or family history of congenital long QT syndrome
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator
* History of GI surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that uncomplicated appendectomy and hernia repair will be allowed
* History of myocardial infarction
* History of febrile illness within 10 days prior to the first dose of study drug, or participants with evidence of active systemic infection, as determined by the investigator
* History of acute GI symptoms (e.g., nausea, vomiting, diarrhea, heartburn) as determined by the investigator (or designee) at Screening or Check-in
* History of ophthalmological disease or clinically significant abnormality in the ophthalmic examination as determined by the investigator, optometrist, or ophthalmologist
* Risk for suicidal behavior at Screening as determined by the investigator's clinical assessment and an answer "Yes" to item 4 or 5 within 2 years of Screening, or to suicidal behavior items on the Baseline/Screening version C-SSRS or suicide attempt within 2 years of screening. Non-suicidal self-injurious behavior is not exclusionary.
* Have significantly impaired hepatic function (at Screening or Check-in)
* Female who is pregnant or breastfeeding or intending to become pregnant during the study or within 90 days following the final ZN-A-1041 administration
* Have a corrected QT (QTc) interval corrected through use of Fredericia's formula >450 msec for males or >470 for females, PR interval >210 msec, QRS complex >120 msec, or heart rate <50 bpm (at Screening or Check-in)
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically significant, such as symptomatic bradyarrhythmias, bradycardia, or heart block as determined from 12-lead ECG (at Screening, Check-in, or Day 1 predose). Abnormal results can be confirmed by one repeat 12-lead ECG
* History of alcoholism or drug addiction within 1 year prior to Check-in, use of drugs of abuse (including opioids) within 4 weeks of Screening, and/or positive alcohol breath test and/or urinary drug screen at Screening or Check-in
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 90 days, whichever is longer, prior to Check-in
* Treatment with intravenous (IV) antibiotics within 8 weeks prior to Screening and/or treatment with oral antibiotics within 4 weeks prior to Screening
* Use of any drugs known to be moderate or strong inhibitors or inducers of CYP3A or CYP2C8 within 30 days prior to Check-in
* Use of any other prescription medications/products or vaccines (including seasonal flu, H1N1, and coronavirus 2019 [COVID-19] vaccines) other than oral, implantable, transdermal, and injectable contraceptives or medications administered during the ophthalmic examination within 14 days prior to Check-in, unless deemed acceptable by the investigator
* Use of therapeutic anticoagulation or thrombolytic anticoagulants within 14 days prior to Check-in
* Use of any over-the-counter, non-prescription medications (including vitamins; minerals; and phytotherapeutic-, herbal-, and plant-derived preparations) within 7 days prior to Check-in, unless deemed acceptable by the investigator
* Use of tobacco- or nicotine-containing products (including, but not limited to, cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 3 months prior to Check-in or a positive cotinine test
* Use of poppy seed-, grapefruit-, star fruit-, pomegranate-, pawpaw-, or Seville orange-containing foods or beverages within 7 days prior to Check-in
* Use of alcohol- or caffeine-containing foods or beverages within 48 hours prior to Check-in, unless deemed acceptable by the investigator
* Participant is not willing to minimize or avoid exposure to natural or artificial sunlight (tanning beds or ultraviolet (UV) A/B treatment) following administration of study drug through 5 days following the final ZN-A-1041 administration
* Participant is not willing to refrain from strenuous exercise from 7 days prior to Check-in and during the period of confinement at the study site (e.g., will not begin a new exercise program or participate in any unusually strenuous physical exertion)
* Poor peripheral venous access as determined by the investigator
* History of malignancy within 5 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix or basal cell skin cancer)
* Donation of blood within 3 months prior to Screening through study completion, donation of plasma within 2 weeks prior to Screening through study completion, or donation of platelets within 6 weeks prior to Screening through study completion
* Receipt of blood products within 2 months prior to Screening and during the entire study duration
* Participants who, in the opinion of the investigator (or designee), should not participate in this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) | Days 1 to 8, 11 to 14, and 17 to 20
Area Under the Concentration-time Curve (AUC) From Hour 0 to the Last Measurable Concentration (AUC0-t) | Days 1 to 8, 11 to 14, and 17 to 20
AUC Extrapolated to Infinity (AUC0-∞) | Days 1 to 8, 11 to 14, and 17 to 20
Geometric Mean Ratio and Associated 90% Confidence Interval (CI) of Cmax, AUC0-t, and AUC0-∞ | Days 1 to 8, 11 to 14, and 17 to 20

SECONDARY OUTCOMES:
ZN-A-1041 PK Parameters Time to Maximum Observed Concentration (Tmax) for All Treatments | Days 1 to 8, 11 to 14, and 17 to 20
ZN-A-1041 Apparent Terminal Elimination Rate Constant (λz) for All Treatments | Days 1 to 8, 11 to 14, and 17 to 20
ZN-A-1041 Apparent Terminal Elimination Half-life (t1/2) for All Treatments | Days 1 to 8, 11 to 14, and 17 to 20
ZN-A-1041 Apparent Systemic Clearance (CL/F) for All Treatments | Days 1 to 8, 11 to 14, and 17 to 20
ZN-A-1041 Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) for All Treatments | Days 1 to 8, 11 to 14, and 17 to 20
Incidence of Adverse Events (AEs), Including Serious Adverse Events (SAEs) and AEs of Special Interest (AESIs) | Up to approximately 8.5 weeks
Severity of AEs, Including SAEs and AESIs | Up to approximately 8.5 weeks
Number of Participants with Abnormalities in Clinical Laboratory Results | Baseline, Days 2, 4, 6, 10, 16, and 20
Changes from Baseline in Oral Temperature Measurements | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20
Columbia Suicide Severity Rating Scale (C-SSRS) Questionnaires | Baseline, Day 1, 5, 11, 17, and 20
Changes from Baseline in Respiratory Rate Measurements | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20
Changes from Baseline in Systolic Blood Pressure Measurements | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20
Changes from Baseline in Pulse Rate Measurements | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20
Changes from Baseline in Diastolic Blood Pressure Measurements | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20
Changes from Baseline in 12-lead Electrocardiogram (ECG) Parameters (RR, PR, QRS, and QT Duration) | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20
Changes from Baseline in 12-lead ECG Parameters (Heart Rate) | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20
Changes from Baseline in 12-lead ECG Parameters (Sinus Rhythm) | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20
Changes from Baseline in 12-lead ECG Parameters (QTcF) | Baseline, Days 1, 2, 5, 6, 11, 12, 17, 18, and 20

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Daytona Beach Clinical Rsch Unit, Daytona Beach, Florida
  - Fortrea Clinical Research Unit - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No